CLINICAL TRIAL: NCT05668741
Title: A Phase 1/2 Dose Escalation Study Evaluating the Safety, and Tolerability and Efficacy of VX-522 in Subjects 18 Years of Age and Older With Cystic Fibrosis and a CFTR Genotype Not Responsive to CFTR Modulator Therapy
Brief Title: A Phase 1/2 Study of VX-522 in Participants With Cystic Fibrosis (CF)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Moderna, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX21-522-001; 2022-000726-25 (EudraCT Number); 2023-504786-23-00 (Other: EU CT Number)
Record Dates: First submitted 2022-12-19; First posted 2022-12-30 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose (SAD) (Experimental): Participants grouped into different cohorts will receive a single ascending dose of VX-522.
  Interventions: Drug: VX-522 mRNA therapy
- Multiple Ascending Dose (MAD) Cohort 1: VX-522 (Experimental): Participants will receive multiple ascending doses of VX-522.
  Interventions: Drug: VX-522 mRNA therapy
- MAD Cohort 1: VX-522+ IVA (Experimental): Following run-in period with ivacaftor (IVA), participants will receive multiple ascending doses of VX-522 with IVA.
  Interventions: Drug: VX-522 mRNA therapy; Drug: IVA
- MAD Cohort 2: VX-522+ IVA (Experimental): Following run-in period with ivacaftor (IVA), participants will receive multiple ascending doses of VX-522 with IVA.
  Interventions: Drug: VX-522 mRNA therapy; Drug: IVA

INTERVENTIONS:
Drug: VX-522 mRNA therapy — Oral inhalation using nebulizer.
Drug: IVA — Tablet for oral administration.
  Other Names: ivacaftor; VX-770
  Arms: MAD Cohort 1: VX-522+ IVA; MAD Cohort 2: VX-522+ IVA

SUMMARY:
The purpose of this study is to evaluate the safety, and tolerability and efficacy of VX-522 in participants 18 years of age and older with cystic fibrosis and a cystic fibrosis transmembrane conductance regulator (CFTR) genotype not responsive to CFTR modulator therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index is less than (<) 30.0 kilograms per meter square (kg/m^2)
* A total body weight greater than (>) 50 kg
* Stable CF disease
* CFTR gene mutations on both alleles that are not responsive to CFTR modulator therapy

  o Example mutations include but are not limited to, mutations that do not produce CFTR protein (i.e., Class I): nonsense mutations (e.g., G542X, W1282X) and canonical splice mutations (e.g., 621+1G->T)
* Forced expiratory volume in 1 second (FEV1) value for SAD: greater than or equal to (≥)40 percent (%), MAD: ≥ 40% to less than or equal to (≤) 90%

Key Exclusion Criteria:

* History of uncontrolled asthma within a year prior to screening
* History of solid organ or hematological transplantation
* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment (Child Pugh Score 7 to 9), or severe hepatic impairment (Child Pugh Score 10 to 15)
* Arterial oxygen saturation on room air less than (<) 94% at screening

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2026-12-23 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 Through Week 8 [SAD and MAD]

SECONDARY OUTCOMES:
MAD: Change From Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) | From Baseline at Day 29
MAD: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 Through Safety Follow-up Visit [up to Week 28]

CONTACTS AND LOCATIONS:
Locations (43):
- United States (24):
  - University of Alabama at Birmingham - Child Health Research Unit, Birmingham, Alabama
  - Memorial Health Services on behalf of Long Beach Memorial Medical Center d/b/a Miller Children's Hospital Long Beach, Long Beach, California
  - Stanford University - Palo Alto - Pulmonology, Palo Alto, California
  - National Jewish Health, Denver, Colorado
  - Shands Hospital - Pulmonology, Gainesville, Florida
  - Northwestern Memorial Hospital - Feinberg Pavilion, Chicago, Illinois
  - Clinical & Translational Science Unit (CTSU) - Pulmonology, Kansas City, Kansas
  - PAREXEL International - Baltimore, Baltimore, Maryland
  - The Johns Hopkins University - Johns Hopkins Hospital - Pulmonology, Baltimore, Maryland
  - MGH - MGfC Pediatric Cystic Fibrosis Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota -Pulmonology, Minneapolis, Minnesota
  - St. Louis Children's Hospital - Pulmonology, St Louis, Missouri
  - Medicine at East 85th Street, New York, New York
  - Presbyterian Hospital - Pulmonology, New York, New York
  - UC Health Holmes Hospital, Cincinnati, Ohio
  - UH Cleveland Medical Center - Pulmonology, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh - Pulmonology, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Pulmonology, Charleston, South Carolina
  - Vanderbilt Interventional Pulmonology, Nashville, Tennessee
  - Texas Children's Hospital - Wallace Tower - Pulmonology, Houston, Texas
  - University of Utah Hospital - Pulmonology, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- The Alfred Hospital - Pulmonology, Melbourne, Australia
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Canada (2):
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - IUCPQ Pavillon Recherche U-1771, Québec
- Ruhrlandklinik, Essen, Germany
- Italy (3):
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico - Pulmonology, Genova
  - IRCSS Ospedale Pediatrico Bambino Gesu - Pulmonology, Rome
  - Centro Ricerche Cliniche di Verona S.r.l., Verona
- UMCU - Department of Pulmonology and Tuberculosis, Utrecht, Netherlands
- Spain (3):
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Virgen del Rocio - Pulmonology, Seville
  - Hospital Universitario y Politecnico La Fe - Pulmonology, Valencia
- Karolinska University Hospital - Pulmonology, Stockholm, Sweden
- United Kingdom (6):
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Queen Elizabeth University Hospital - Pulmonology, Glasgow
  - Royal Brompton Hospital, London
  - Wythenshawe Hospital - OPD, Manchester
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth
  - University Hospital Southampton NHS Fountion - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/